CLINICAL TRIAL: NCT02924454
Title: An Investigation Into the Effects of Intravenous Lipid Emulsion (ILE) on the Pharmacokinetic and Pharmacodynamic Properties of Metoprolol.
Brief Title: Effects of Lipid Emulsion on the Pharmacokinetic and Pharmacodynamic Properties of Metoprolol.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mikkel Bring Christensen (Other)
Responsible Party: Sponsor-Investigator, Mikkel Bring Christensen, MD, PhD, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Intralipid-Metoprolol
Record Dates: First submitted 2016-09-06; First posted 2016-10-05 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Drug Overdose; Overdose of Beta-adrenergic Blocking Drug; Blood Pressure
Keywords: metoprolol; lipid emulsion; pharmacodynamics; pharmacokinetics
MeSH Terms: conditions — Drug Overdose | interventions — Metoprolol; Fat Emulsions, Intravenous; soybean oil, phospholipid emulsion; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Metoprolol-Lipid emulsion (Experimental): intervention 1: metoprolol Intervention 2: intravenous lipid emulsion
  Interventions: Drug: metoprolol; Drug: intravenous lipid emulsion
- Metoprolol - normal saline (Experimental): intervention 1: metoprolol intervention 2: Sodium chloride 0.9% solution - lipid emulsion dummy
  Interventions: Drug: metoprolol; Drug: Sodium chloride 0.9% solution - lipid emulsion dummy
- Normal saline-Lipid emulsion (Experimental): intervention 1: Sodium chloride 0.9% solution - metoprolol dummy intervention 2: intravenous lipid emulsion
  Interventions: Drug: intravenous lipid emulsion; Drug: Sodium chloride 0.9% solution - metoprolol dummy
- Normal saline-normal saline (Experimental): intervention 1: Sodium chloride 0.9% solution - metoprolol dummy intervention 2: Sodium chloride 0.9% solution - lipid emulsion dummy
  Interventions: Drug: Sodium chloride 0.9% solution - lipid emulsion dummy; Drug: Sodium chloride 0.9% solution - metoprolol dummy

INTERVENTIONS:
Drug: metoprolol — One hundred and twenty ml, 0.5 mg metoprolol/ml (as metoprolol tartrate) is administered as an intravenous bolus injection followed by a continuous infusion. Infusion is halted if heart rate drops below 35 bpm or systolic blood pressure drops below 80 mm Hg, or the participant experiences subjective side effects. Infusion stops at T=30 minutes.
  Other Names: metoprolol tartrate; Seloken; ATC: C07AB02
  Arms: Metoprolol - normal saline; Metoprolol-Lipid emulsion
Drug: intravenous lipid emulsion — Intravenous lipid emulsion 20 % is administered as an intravenous bolus infusion (1.5 ml/kg) followed by continuous infusion (infusion rate: 0.25 ml/kg/min). Lipid emulsion infusion is stopped at T = 30 minutes.
  Other Names: Intralipid; ATC: B05BA02
  Arms: Metoprolol-Lipid emulsion; Normal saline-Lipid emulsion
Drug: Sodium chloride 0.9% solution - lipid emulsion dummy — Isotonic 0.9 % sodium chloride solution is administered as an intravenous bolus infusion (1.5 ml/kg), followed by continuous infusion (infusion rate: 0.25 ml/kg/min). Infusion is stopped at T = 30 minutes.
  Other Names: Normal saline
  Arms: Metoprolol - normal saline; Normal saline-normal saline
Drug: Sodium chloride 0.9% solution - metoprolol dummy — Saline solution is administered as an intravenous bolus injection followed by a continuous infusion to T=30 minutes.
  Other Names: Normal saline
  Arms: Normal saline-Lipid emulsion; Normal saline-normal saline

SUMMARY:
The aim of this study is to investigate whether intravenous lipid emulsion is effective in attenuating the clinical effects of a cardioactive drug, exemplified by the beta-blocking agent metoprolol. In addition, the investigators will clarify how intravenous lipid emulsion affects the pharmacokinetic parameters of metoprolol.

DETAILED DESCRIPTION:
Overdose or poisonings with cardioactive drugs can have serious consequences. In recent years, intravenous lipid emulsion has emerged as a possible treatment option in otherwise treatment-resistant cardiovascular collapse caused by poisonings with cardio-active drugs.

Experimental evidence obtained from animal studies has been indicating a beneficial effect of intravenous lipid emulsion in the treatment of poisoning with various cardio-toxic medications. Based on these findings, the first reported cases on the use of intravenous lipid emulsion in the treatment of human cardiotoxicity caused by poisonings with local anesthetics were published in 2006. Subsequently, a steadily increasing number of case reports concerning the use of intravenous lipid emulsion in resuscitation and treatment of various medications poisonings have been published. Often patients had either cardiac arrest or severe circulatory failure treated according to guidelines for advanced life support prior to lipid emulsion therapy. It is noteworthy that a common observation following bolus infusion of lipid emulsion has been a rapid hemodynamic stabilization of the patient.

Despite an increasing use of intravenous lipid emulsion in the treatment of the poisoned patient, the mechanism behind lipid rescue has not been elucidated. The most widely accepted hypothesis, the "lipid sink/sponge" model, suggests that intravenous lipid emulsion entraps xenobiotics intravascularly, thereby preventing them from reaching sites of toxicity. Additionally, intravenous lipid emulsion may redistribute xenobiotics to areas of higher lipid content. However, other mechanisms of actions of lipid emulsion, supported by observations from animal experiments, are vasoconstrictive and cardio-tonic effects. These effects could be secondary to direct activation of sodium, potassium or calcium channels in the myocardium, or alternatively fatty acid-induced modulation of the metabolic properties of mitochondria. Both mechanisms could result in hemodynamic stabilization. The potential beneficial effects of lipid emulsion on hemodynamic instability beyond the lipid sink have led to the notion that intravenous lipid emulsion could be valuable in the treatment of poisonings with non-lipophilic xenobiotics.

At present, it remains however unclear to what extent the evidence concerning resuscitation of the poisoned patient with lipid emulsion may reflect publication bias. To our knowledge, only one controlled human trial has been conducted at present. In a randomized crossover study, Litonius et al. investigated the effects of lipid emulsion on plasma concentrations of bupivacaine in eight healthy subjects. It was found that lipid emulsion lowered the total plasma concentrations of bupivacaine. This was attributed to an altered distribution and contradicted so the above hypothesis of a lipid sink-mechanism as the fraction of non-lipid bound bupivacaine was unchanged. The mechanism by which lipid emulsion may attenuate the effects of cardio toxic xenobiotics must therefore still be regarded as undecided. This lack of evidence calls for further human studies in order to elucidate the pharmacokinetic and pharmacodynamic consequences of intravenous lipid emulsion. The purpose of this double blind, randomized placebo-controlled crossover clinical trial is to investigate the effects of intravenous lipid emulsion on the pharmacokinetic and pharmacodynamic properties of the adrenoceptor antagonist metoprolol in a human model of beta blocker overdose.

The study includes a total of five visits; a screening visit and four trial days. At the screening visit, anthropometric data (weight, height, blood pressure and pulse) is measured. Additionally, blood samples are collected in accordance with exclusion criteria. A spot urine sample measuring the albumin/creatinine ratio is collected and an electrocardiogram (ECG) is recorded to verify normality of heart rhythm and electrical impulses. In addition, an investigator carries out a clinical examination. Based on the clinical examination, urine and blood tests and ECG measurement, the investigator assesses whether the trial participant meet all inclusion criteria and no exclusion criteria.

After screening and inclusion, participants will be invited to four trial days at the trial site. On each day participants are required to be fasting for 10 hours (including water, coffee and tobacco). A peripheral venous line is inserted into each antecubital vein. An arterial catheter connected to a pressure transducer is inserted into the radial artery in the wrist. In randomized order, one of the four interventions are performed (see below). A standard 12 lead ECG is placed on the participant as well as a 5 lead ECG connected to a computer.

At T=0, metoprolol intravenous solution (0.5 mg metoprolol/ml as metoprolol tartrate) or placebo is administered as an intravenous bolus injection. Continuous infusion of metoprolol/placebo is then administered until T=30 minutes. Infusion is halted if heart rate drops below 35 bpm or systolic blood pressure drops below 80 mm Hg, or the participant experiences subjective side effects. Infusion stops at T=30 minutes. Intravenous lipid emulsion (Intralipid 20 %) or saline solution is shortly thereafter administered as an intravenous bolus infusion (1.5 ml/kg) followed by a continuous infusion (infusion rate: 0.25 ml/kg/min). Lipid emulsion/dummy infusion is stopped at T = 30 minutes. One gram of paracetamol administered as a disintegrating tablet dissolved in 50 ml of water is given per os shortly before study start on each day.

Repeated ECG's are recorded and blood is drawn for measurements of routine biochemistry parameters and serum concentrations of metoprolol and paracetamol. A drop of blood is used to test glucose levels using a blood glucose meter. Cardiovascular parameters (heart rate, blood pressure, pulse contour curve/arterial pressure wave) are recorded via the arterial catheter and pressure transducer connected to a computer. The participant is closely monitored on site until T=120 minutes.

ELIGIBILITY:
Inclusion Criteria:

- healthy male.

Exclusion Criteria:

* Abnormal blood levels of sodium, potassium, creatinine, alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase, albumin, bilirubin, hemoglobin, HbA1c, cholesterol fractions.
* Abnormal urine albumin to creatinine ratio.
* Abnormal function of CYP2D6 metabolism (ultrarapid or slow metabolizer)
* Any heart disease or hypertension
* Sinoatrial block
* Second or third degree atrioventricular block
* Heart failure
* profound bradycardia or hypotension
* sinoatrial node disease
* metabolic acidosis
* untreated pheochromocytoma
* asthma
* chronic obstructive pulmonary disease
* intermittent claudicatio
* diabetes
* Allergy to egg, soy or peanut protein and allergy to any active or inactive ingredients contained in metoprolol (Seloken) or the lipid emulsion (Intralipid)
* Raynaud's syndrome
* Prinzmetal's angina

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Change in heart rate from baseline compared between study days | From baseline to + 120 minutes.
  Arterial catheter connected to a pressure transducer records heart rate (beats per minute).

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of metoprolol on days with co-administration of intravenous lipid emulsion compared to days with lipid emulsion placebo. | 0, +10, +20, +30, +40, +50, +60, +90, +120 minutes post metoprolol dose.
  Blood samples drawn from an antecubital vein.
Peak plasma concentration (Cmax) of paracetamol on days with co-administration of intravenous lipid emulsion compared to days with lipid emulsion placebo. | 0, +10, +20, +30, +40, +50, +60, +90, +120 minutes post metoprolol dose.
  Paracetamol is used as a tool for measuring gastric emptying time.
Area under the plasma concentration versus time curve (AUC) of paracetamol on days with co-administration of intravenous lipid emulsion compared to days with lipid emulsion placebo. | 0, +10, +20, +30, +40, +50, +60, +90, +120 minutes post metoprolol dose.
  Paracetamol is used as a tool for measuring gastric emptying time.
Time to peak plasma concentration (Tmax) of paracetamol on days with co-administration of intravenous lipid emulsion compared to days with lipid emulsion placebo. | 0, +10, +20, +30, +40, +50, +60, +90, +120 minutes post metoprolol dose.
  Paracetamol is used as a tool for measuring gastric emptying time.
Percent change in plasma levels of standard biochemical measurements from baseline compared between study days. | Changes at +30 and +60 minutes from baseline.
  Blood samples drawn from an antecubital vein measuring alanine aminotransferase, aspartate aminotransferase, albumin, bilirubin, alkaline phosphatase, calcium, creatine kinase, creatinine, C-reactive protein, high density lipoprotein, potassium, sodium, glucagon, lactate dehydrogenase, haptoglobin, triglycerides, and whole blood glucose levels(measured with a glucose meter).
Peak Plasma Concentration (Cmax) of metoprolol on days with co-administration of intravenous lipid emulsion compared to days with lipid emulsion placebo. | +0, +10, +20, +30, +40, +50, +60, +90, +120 minutes post metoprolol dose.
  Blood samples drawn from an antecubital vein measuring plasma metoprolol.
Time to peak plasma concentration (Tmax) of metoprolol on days with co-administration of intravenous lipid emulsion compared to days with lipid emulsion placebo. | +0, +10, +20, +30, +40, +50, +60, +90, +120 minutes post metoprolol dose.
  Blood samples drawn from an antecubital vein measuring plasma metoprolol.
Cardiac conductivity between days with metoprolol and/or intravenous lipid emulsion compared with placebo. | T-10, T-5, T 0, T 10, T 20, T 30, T 40, T 50, T 60, T 90, T 120 minutes.
  12-lead ECG
Effects of metoprolol and lipid emulsion on stroke volume compared to days with placebo. | T-10, T-5, T 0, T 10, T 20, T 30, T 40, T 50, T 60, T 90, T 120 minutes.
  Stroke volume (mL) derived from arterial pulse contour analysis.
Effect of metoprolol on systolic, diastolic and mean arterial pressure on days with co-administration of intravenous lipid emulsion compared to days with placebo. | T-10, T-5, T 0, T 10, T 15, T 20, T 30, T 40, T 50, T 60, T 90, T100, T110, T 120 minutes.
  Arterial catheter connected to a pressure transducer records blood pressure in mm Hg.
Change in systolic, diastolic and mean arterial pressure from baseline compared between study days. | Changes at +5, +10, +15, +20, +30, +40, +50, +60, +90, +95, +100, +105, +110, +115, +120 minutes from baseline.
  Arterial catheter connected to a pressure transducer records blood pressure in mm Hg.
Change in heart rate from baseline compared between study days. | Changes at +5, +10, +15, +20, +30, +40, +50, +60, +90, +95, +100, +105, +110, +115, +120 minutes from baseline.
  Arterial catheter connected to a pressure transducer records heart rate (beats per minute).
Change in stroke volume (ml) from baseline compared between study days. | Changes at +5, +10, +15, +20, +30, +40, +50, +60, +90, +95, +100, +105, +110, +115, +120 minutes from baseline.
  Stroke volume (ml) derived from arterial pulse contour analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel B Christensen, MD, PhD, Principal Investigator — Bispebjerg University Hospital, Copenhagen
Locations (1):
- Bispebjerg University Hospital Copenhagen, Copenhagen Northwest, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffman RS, Howland MA, Lewin NA, Nelson L, Goldfrank LR, Flomenbaum N, editors. Goldfrank's toxicologic emergencies. Tenth edition. New York: McGraw-Hill Education; 2015. 1882 p.
- [Background] Picard J, Ward SC, Zumpe R, Meek T, Barlow J, Harrop-Griffiths W. Guidelines and the adoption of 'lipid rescue' therapy for local anaesthetic toxicity. Anaesthesia. 2009 Feb;64(2):122-5. doi: 10.1111/j.1365-2044.2008.05816.x. PMID 19143686
- [Background] Tebbutt S, Harvey M, Nicholson T, Cave G. Intralipid prolongs survival in a rat model of verapamil toxicity. Acad Emerg Med. 2006 Feb;13(2):134-9. doi: 10.1197/j.aem.2005.08.016. Epub 2006 Jan 25. PMID 16436797
- [Background] Di Gregorio G, Schwartz D, Ripper R, Kelly K, Feinstein DL, Minshall RD, Massad M, Ori C, Weinberg GL. Lipid emulsion is superior to vasopressin in a rodent model of resuscitation from toxin-induced cardiac arrest. Crit Care Med. 2009 Mar;37(3):993-9. doi: 10.1097/CCM.0b013e3181961a12. PMID 19237909
- [Background] Weinberg G, Ripper R, Feinstein DL, Hoffman W. Lipid emulsion infusion rescues dogs from bupivacaine-induced cardiac toxicity. Reg Anesth Pain Med. 2003 May-Jun;28(3):198-202. doi: 10.1053/rapm.2003.50041. PMID 12772136
- [Background] Weinberg GL, Di Gregorio G, Ripper R, Kelly K, Massad M, Edelman L, Schwartz D, Shah N, Zheng S, Feinstein DL. Resuscitation with lipid versus epinephrine in a rat model of bupivacaine overdose. Anesthesiology. 2008 May;108(5):907-13. doi: 10.1097/ALN.0b013e31816d91d2. PMID 18431127
- [Background] Weinberg GL, VadeBoncouer T, Ramaraju GA, Garcia-Amaro MF, Cwik MJ. Pretreatment or resuscitation with a lipid infusion shifts the dose-response to bupivacaine-induced asystole in rats. Anesthesiology. 1998 Apr;88(4):1071-5. doi: 10.1097/00000542-199804000-00028. PMID 9579517
- [Background] Rosenblatt MA, Abel M, Fischer GW, Itzkovich CJ, Eisenkraft JB. Successful use of a 20% lipid emulsion to resuscitate a patient after a presumed bupivacaine-related cardiac arrest. Anesthesiology. 2006 Jul;105(1):217-8. doi: 10.1097/00000542-200607000-00033. No abstract available. PMID 16810015
- [Background] Litz RJ, Popp M, Stehr SN, Koch T. Successful resuscitation of a patient with ropivacaine-induced asystole after axillary plexus block using lipid infusion. Anaesthesia. 2006 Aug;61(8):800-1. doi: 10.1111/j.1365-2044.2006.04740.x. PMID 16867094
- [Background] Bet 2: intralipid/lipid emulsion in beta-blocker overdose. Emerg Med J. 2011 Nov;28(11):991-3. doi: 10.1136/emermed-2011-200722. PMID 22002529
- [Background] Blaber MS, Khan JN, Brebner JA, McColm R. "Lipid rescue" for tricyclic antidepressant cardiotoxicity. J Emerg Med. 2012 Sep;43(3):465-7. doi: 10.1016/j.jemermed.2011.09.010. Epub 2012 Jan 12. PMID 22244291
- [Background] Espinet AJ, Emmerton MT. The successful use of intralipid for treatment of local anesthetic-induced central nervous system toxicity: Some considerations for administration of intralipid in an emergency. Clin J Pain. 2009 Nov-Dec;25(9):808-9. doi: 10.1097/AJP.0b013e3181af739e. PMID 19851162
- [Background] Finn SD, Uncles DR, Willers J, Sable N. Early treatment of a quetiapine and sertraline overdose with Intralipid. Anaesthesia. 2009 Feb;64(2):191-4. doi: 10.1111/j.1365-2044.2008.05744.x. PMID 19143698
- [Background] Foxall G, McCahon R, Lamb J, Hardman JG, Bedforth NM. Levobupivacaine-induced seizures and cardiovascular collapse treated with Intralipid. Anaesthesia. 2007 May;62(5):516-8. doi: 10.1111/j.1365-2044.2007.05065.x. PMID 17448066
- [Background] Ludot H, Tharin JY, Belouadah M, Mazoit JX, Malinovsky JM. Successful resuscitation after ropivacaine and lidocaine-induced ventricular arrhythmia following posterior lumbar plexus block in a child. Anesth Analg. 2008 May;106(5):1572-4, table of contents. doi: 10.1213/01.ane.0000286176.55971.f0. PMID 18420879
- [Background] Marwick PC, Levin AI, Coetzee AR. Recurrence of cardiotoxicity after lipid rescue from bupivacaine-induced cardiac arrest. Anesth Analg. 2009 Apr;108(4):1344-6. doi: 10.1213/ane.0b013e3181979e17. PMID 19299810
- [Background] Shah S, Gopalakrishnan S, Apuya J, Shah S, Martin T. Use of Intralipid in an infant with impending cardiovascular collapse due to local anesthetic toxicity. J Anesth. 2009;23(3):439-41. doi: 10.1007/s00540-009-0754-3. Epub 2009 Aug 14. PMID 19685131
- [Background] Warren JA, Thoma RB, Georgescu A, Shah SJ. Intravenous lipid infusion in the successful resuscitation of local anesthetic-induced cardiovascular collapse after supraclavicular brachial plexus block. Anesth Analg. 2008 May;106(5):1578-80, table of contents. doi: 10.1213/01.ane.0000281434.80883.88. PMID 18420881
- [Background] Weinberg GL. Lipid infusion therapy: translation to clinical practice. Anesth Analg. 2008 May;106(5):1340-2. doi: 10.1213/ane.0b013e31816a6c09. No abstract available. PMID 18420841
- [Background] Fettiplace MR, Akpa BS, Ripper R, Zider B, Lang J, Rubinstein I, Weinberg G. Resuscitation with lipid emulsion: dose-dependent recovery from cardiac pharmacotoxicity requires a cardiotonic effect. Anesthesiology. 2014 Apr;120(4):915-25. doi: 10.1097/ALN.0000000000000142. PMID 24496123
- [Background] Litonius E, Tarkkila P, Neuvonen PJ, Rosenberg PH. Effect of intravenous lipid emulsion on bupivacaine plasma concentration in humans. Anaesthesia. 2012 Jun;67(6):600-5. doi: 10.1111/j.1365-2044.2012.07056.x. Epub 2012 Feb 21. PMID 22352703